CLINICAL TRIAL: NCT06403059
Title: Cervical Length and Uterocervical Angle as Predictors of Spontaneous Preterm Birth
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: CL in preterm
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Preterm Pregnancy
Keywords: preterm delivery; Cervical Length; Uterocervical Angle
MeSH Terms: conditions — Premature Birth | interventions — Cervical Length Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cervical Length — trans vaginal ultrasound
Diagnostic Test: Uterocervical Angle — by trans vaginal ultrasound

SUMMARY:
This prospective study was carried out on 263 pregnant females aged from 19 to 35 years old carrying singleton, and uncomplicated pregnancy. TVS examination was performed in all cases at 28 and 32 weeks of gestation. The pregnant women recruited in the study closely followed up to delivery. Maternal progesterone was given to all women with short CL (<20mm and more than 10mm) to support pregnancy.

DETAILED DESCRIPTION:
#Patients and Methods: This prospective cohort study was performed on 263 pregnant females aged from 19 to 35 years old carrying singleton, and uncomplicated pregnancy.

The study was done after approval from ethical committee. An informed written consent was obtained from the patient.

With aseptic measures and a high-frequency endo-vaginal 7.5 Hz. probe (GE Logiq P6), TVS examinations were done to all pregnant women. Dorsal lithotomy posture was applied to pregnant women who were instructed to evacuate their bladders. Without applying excessive pressure, the vaginal probe was inserted into the anterior fornix. At maximum magnification, a sagittal image of the cervix and anterior uterine wall was obtained. We identified the echogenic endocervical canal with the surrounded less echogenic cervical mucosa zone. The external os was noted at the junction of the cervix both anterior and posterior lips within the vaginal canal, but the internal os was situated at the end of the cervical mucosa in the lower uterine segment. CL and UCA were measured using the ultrasound's built-in angle caliper. The anterior UCA measurement involved calculating the angle formed by a line running through the cervix and another line along the lower front segment of the uterus, starting from the internal os. This was achieved by manually drawing two lines with the angle caliper: one connecting the internal and external os, and another extending from the internal os along the lower anterior uterine wall, up to a point 3 cm from the internal os.

The research involved close monitoring of pregnant participants up to the time of delivery. Demographics and pregnancy outcomes were collected and recorded. PTB was defined as delivery occurring before 37 complete weeks of gestation [9]. To support pregnancy, maternal progesterone was administered to all women with a short CL (less than 20mm but more than 10mm). In this study, cervical cerclage was not used in any case.

Sample Size Calculation:

The sample size for the study was determined using the Open-Epi, Version 3, an open-source software tool. This calculation was based on the premise that 78.1% of patients with a cervical angle greater than 95 degrees experience preterm labor. To ensure a confidence level of 95% and a margin of error of 5%, it was necessary to include at least 263 patients in the study. The confidence limits were set at 5%, and the design effect was established at 1. The formula used for this calculation was: n = [DEFFNp(1-p)]/ [(d²/Z²1-α/2(N-1) +p*(1-p)].

Statistical analysis Statistical analysis was done by SPSS v26 (IBM Inc., Chicago, IL, USA). Quantitative variables were presented as mean and standard deviation (SD). Qualitative variables were presented as frequency and percentage (%). Correlation between various variables was done using Pearson coefficient. The diagnostic performance was assessed using ROC curve analysis, with the AUC serving as a predictor of sPTB.

ELIGIBILITY:
Inclusion Criteria:

* pregnant 28 to 32 weeks

Exclusion Criteria:

* additional signs of preterm labour in the mother
* foetus, polyhydramnios,
* multiple pregnancies,
* a previous cervix operation,

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 28 to 32 weeks
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
cervical length | 28 and 32 weeks of gestation
  TVS examination
uterocervical angle | 28 and 32 weeks of gestation
  TVS examination

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided